CLINICAL TRIAL: NCT06640270
Title: Evaluation of the PERFormances of a Bioelectrical Impedancemetry Device (Lucie™), for the Measurement of Hydration Parameters in Patients with Renal Failure: a Multicentre Comparative Study
Brief Title: Performance Evaluation of Lucie™ for Hydration of Dialysis Patients
Acronym: PERF-LUCIE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Home Habilis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: PERF-LUCIE
Record Dates: First submitted 2024-09-26; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Diabetes
Keywords: bioimpedance; concordance; hydration match; overhydration; Total Body Water; Extra Cellular Water; Intra Cellular Water; hydration; Over Hydration; predictive value
MeSH Terms: conditions — Diabetes Mellitus; Water Intoxication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Main Arm for PREF-Lucie (Experimental): Interventional, quasi-experimental, multicentre, comparative clinical research study
  Interventions: Device: Diabetes Treatment

INTERVENTIONS:
Device: Diabetes Treatment — Lucie™ is an innovative medical device for measurement by bio-impedancemetry. It has been developed specifically to meet medical needs in nephrology. The aim of the study is to compare its performance with a reference device validated in nephrology nephrology, the Body Composition Monitor® (BCM) from Fresenius.

SUMMARY:
The main objective of the observatory study is to evaluate the performance of the Lucie™ medical device for measuring water balance before and after dialysis (water overload, dry weight) in patients with chronic renal failure. We will compare the results and performance of the device with the reference device in nephrology: the BCM®. This comparison is based on bioimpedance. Bioimpedance is an effective technology for monitoring hydration if used regularly, and will give you greater autonomy in your home monitoring. It competes with other technologies that we have found to be less effective. This is what clinical research is seeking to demonstrate: only a clinical study can verify the reliability of this hypothesis. The aim is to help Lucie technology mature so that it can detect early signs of fluid overload, and ultimately prevent complications or hospitalisation.

The process is as follow:

* After removing their shoes and socks, the patient will be invited to step onto the scale;
* Patient will insert a personal card into the card reader and place his right hand loosely on the LucieTM handle, keeping a natural posture;
* The device will take measurements for 45 seconds under the nurse's supervision;
* Patient will go down Lucie and will answer a short form;
* The device is cleaned after each use For optimum results, we recommand patients to keep their feet dry and their hands clean (without cream), and we recommend them to remove their jewellery, to keep their smartphones away from the device (to avoid interference), and to wear a minimum of nylon-free clothing, with empty pockets.

In practical terms, patients are familiar with monitoring their fluid overload using the Fresinus BCM® bathroom scale. They already use it as part of their clinical routine when entering and leaving the dialysis room. This BCM® is used at the start of the dialysis session, before the session begins, by a nurse trained by the manufacturer in its use: he or she knows how to place the electrodes and read the results for status and fluid overload. The nurse also takes patients' usual vital signs (blood pressure, temperature) and notes any incidents during the dialysis session (low blood pressure, cramps, headaches, nausea, etc.) in line with standard practice.

With Lucie™

DETAILED DESCRIPTION:
The goal of this observational study is to evaluate the performance of the Lucie™ medical device for the measurement of pre-dialytic hyperhydration by bioimpedance (water volume in L) in groups of patients with renal failure, compared with the reference device, the BCM. The main question its aimed to answer is

The primary hypothesis will be to determine the degree of agreement between the BMC measure of pre-dialytic hyperhydration and Lucie&#39;s water balance (volume (L)).

Participants will do the following tasks :

* Patients weigh themselves on entering the dialysis room to find out their total weight and have it checked by the nurse (routine care) with a scale that complies with weighing standard NF EN 45501:2015 and Directive 2014/31/EU;
* Patients weigh themselves with Lucie™ and complete a bio-impedance measurement cycle in 45 seconds (interventional research);
* A nurse measures the blood pressure on the cuff (CE medical mark), standing and lying down, and determines the ultrafiltration for the dialysis session to be entered on the machine (routine care). She records the pre-dialysis information;
* The nurse performs a bio-impedance measurement with the BCM™ reference device from Fresenius Medical Care and records measurements of hyperhydration - or overhydration (OH) -, extracellular water (ECW), total body water (TBW), the ECW/TBW ratio, the E/I ratio (deep breathing test), the OH/ECW ratio (interventional research);
* Patients begin their dialysis session (routine care);
* The nurse records blood pressure, standing and lying down, after the dialysis session and records post-dialysis information and lists any undesirable events during the dialysis session (e.g. cramps, low blood pressure, headaches, etc.);
* Patients are weighed on leaving the dialysis room to check that they are achieving the prescribed target weight (routine care);
* Patients weigh themselves with Lucie™ and complete a cycle of bioimpedance measurements in 45 seconds under the control of a nurse (interventional research).
* Patients weigh themselves a second time with the Lucie™ device and again complete one cycle of bio-impedance measurement in 45 seconds without nurse supervision (interventional research, the aim of which here is to measure inter-operator reliability).
* No bio-impedance measurement by the BCM™ device after the dialysis session given the difficulty of devoting an extra 30 minutes to patients to carry out a second measurement;
* Lucie™ device surfaces are cleaned according to the procedure provided.

ELIGIBILITY:
Inclusion Criteria:

* Patients age : 18 years min
* Weight minor than 125 kg
* must be able to read
* able to get on and off a bathroom scale, with or without assistance;
* Patient able to stand in balance for 45 seconds with support, alone and barefoot.

Exclusion Criteria:

* persons with vulnerabilities : pregnant women, nursing mothers, persons deprived of their liberty, adults under legal protection, persons in emergency situations (art. L. 1121-5 to 8 and L.1122-1-2 of the Public Health Code)
* patient with an open wound on the extremities (palms and soles of the feet in contact with the device);
* Patient with an electronic cardiac implant;
* An amputee, with or without a prosthesis;
* Patients with paralysis, even partial paralysis;
* Patients with a 3-month mean natraemia of less than 130 mmol/L;
* Patients fitted with a metal prosthesis;
* Patients with behavioural problems that prevent them from taking part in the study;
* Patient already included in another interventional research study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-10-15 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Hydratation parameters | Through study completion (2 months)
  Extra Cellular Water (ECW), Total Body Water (TBW), Intra Cellular Water (ICW) ; the agreement of the variation before and after dialysis with Lucie™ of the hydration parameters (ECW, ICW, ECW/ICW, OH/ECW, TBW) and the actual ultrafiltration of the session displayed on the generator (UF). This measure will help to calculate Bioimpedance measure.
Concordance of Hydration parameters (%) | Through study completion (2 months)
  Concordance of hydration parameters (OH/ECW (%) (Over Hydration) to Extra Cellular Water), ECW/ICW (%) (Extra Cellular Water to Intra Cellular Water) between the 2 medical devices (Lucie™ and BCM® reference device), as well as sensitivity, specificity, positive predictive value, negative predictive value by Lucie™ medical device.

SECONDARY OUTCOMES:
Weight Measures | Through study completion (2 months)
  The agreement between the total weight (kg) measured by the reference device and that measured by Lucie
Skin/eat Temperature Agreement | Through study completion (2 months)
  The agreement between the skin temperature (°C) measured by Lucie and the ear temperature measured at the patient's bed ;
Satisfactiory Questionnaire | Through study publication (4 months)
  Patient satisfaction questionnaire to be completed during the dialysis session and at the end of the study by the healthcare professionals who took part.
Medico-economic Impact | From the end of inclusion to one year after CER publication, assessed to 16 months
  Questionnaire on the medico-economic impact of the use of the Lucie™ device to be completed at the end of the study by the healthcare professionals who took part.
Organisational Impact | From the end of inclusion to one year after CER publication, assessed to 16 months
  Questionnaire on the organisational impact of the deployment of the Lucie™ system to be completed at the end of the study by the healthcare professionals who took part.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: General website of the Sponsor — https://www.home-habilis.fr/